CLINICAL TRIAL: NCT03813342
Title: Retraining the Walking Pattern After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Amy J. Bastian, Ph.D., Professor of Neuroscience, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00097573; 2R37NS090610 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-01-23 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Stroke; Hemiparesis
Keywords: stroke; gait training; visual feedback
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: treadmill with multi-dimensional and one-dimensional feedback
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multichannel Visual Feedback (Experimental): Gait training with visual feedback of joint kinematics. The visual feedback will contain information about the lower limb joint angles. We will instruct subjects to use the feedback to reach a target walking pattern. In this arm, subjects will receive 4 channels of visual information, each of which represents a joint angle (right and left hips, right and left knees).
  Interventions: Behavioral: Gait training with visual feedback of joint kinematics
- Single Channel Visual Feedback (Experimental): Gait training with visual feedback of joint kinematics. The visual feedback will contain information about the lower limb joint angles. We will instruct subjects to use the feedback to reach a target walking pattern. In this arm, subjects will receive 1 channel of visual information that encompasses information from 4 lower limb joint angles (right and left hips, right and left knees).
  Interventions: Behavioral: Gait training with visual feedback of joint kinematics

INTERVENTIONS:
Behavioral: Gait training with visual feedback of joint kinematics — Gait training will be accomplished using a Woodway treadmill. The visual feedback will contain information about the real-time lower-limb joint angles. We will instruct participants to use the feedback to reach a target walking pattern.

SUMMARY:
The purpose of the study is to determine the effects of pairing gait training with different forms of visual feedback about leg movements in individual post-stroke to modify/normalize their gait pattern over time.

DETAILED DESCRIPTION:
Stroke often results in functional gait deficits and abnormal gait patterns. Typically, several features of gait are altered (e.g. knee joint movement decreases and step lengths are asymmetric). Data show that walking patterns after neurologic injury can be changed through gait training, but traditional rehabilitation approaches typically focus on changing one feature of gait at a time. However, the investigators have recently shown that in a single session individuals post-stroke are able to learn to change multiple components of this impaired gait pattern at the same time.

To further leverage this ability to learn multiple things at once, the investigators have also studied how different forms of visual feedback about leg movements may best facilitate individuals to make meaningful changes to multiple features of the gait pattern. Specifically, they have studied two forms of visual feedback - 1) multidimensional, with multiple streams of information about leg movements, and 2) one-dimensional, which distills/summarizes multiple pieces of information about the gait pattern into a single source of feedback. They have shown that the one-dimensional summary feedback is more effective to help people learn a new gait pattern that requires changing multiple features of how they are walking. This work has focused on single training sessions in neurologically intact individuals, but the authors would like to study the effects of longer-term training with these different forms of feedback. Therefore, the purpose of this study is to gather preliminary data to inform the design of a clinical trial of gait training to treat walking deficits post-stroke. The investigators will gather data to determine whether training with different forms of visual feedback about leg movements are effective at improving gait patterns post-stroke - and which form of feedback may be more effective.

The investigators will study adults with cerebral damage due to stroke. Subjects with hemiparesis will undergo training 3 times a week for a total of 12 training session. These 12 sessions will be broken into 2 blocks of 6 sessions, with at least a 2 week break in between. In each block, training will occur with one form of visual (multi- or one-dimensional). Participants will complete training with both forms of feedback, the order of feedback forms will be randomly assigned. These studies will provide important new information about gait training with visual feedback in individuals post-stroke. This study is critical for developing procedural reliability processes, calculating effect sizes, and determining other salient clinical variables in preparation for a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* stroke or hemiparesis (>6 months post stroke)
* able to walk but has a residual gait deficit (including those who walk with a cane or walker)
* Able to walk for 5 minutes at their self-paced speed
* Adults age 20-80

Exclusion Criteria:

* Cerebellar signs (e.g.ataxic hemiparesis)
* Any neurologic condition other than stroke
* Uncontrolled diabetes
* Congestive heart failure
* Peripheral artery disease with claudication
* Pulmonary or renal failure
* Unstable angina
* Uncontrolled hypertension (>190/110 mmHg)
* MoCA (Montreal Cognitive Assessment Test for Dementia) < 23
* Severe aphasia
* Orthopedic or pain conditions that limit walking
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
1. Change in hip and knee joint movements while walking | Assessed before and after the gait training provided in each Arm of the study to assess a change following each intervention. This measure will be collected during the first and last sessions of Arms 1 and 2, occurring within two weeks for each Arm.
  How closely the hip and knee movements in participants post-stroke match those of a healthy gait patter. To collect this measure, subjects will wear special markers on their feet and body to record how their legs are moving while they walk on the treadmill.

SECONDARY OUTCOMES:
1. Change in walking speed | Assessed before and after the gait training provided in each Arm of the study to assess a change following each intervention. This measure will be collected during the first and last sessions of Arms 1 and 2, occurring within two weeks for each Arm.
  Subjects will complete clinical tests of walking speed by walking overground at two paces - their normal comfortable pace and as fast as safely possible.
2. Change in subjective assessment of balance confidence | Assessed before and after the gait training provided in each Arm of the study to assess a change following each intervention. This measure will be collected during the first and last sessions of Arms 1 and 2, occurring within two weeks for each Arm.
  Subjects will complete the 16-item Activities-Specific Balance Confidence Scale. This is a self-report measure in which they rate their confidence that they would not lose their balance while performing specific daily activities. Scores can range from 0 - 100, with 0 indicating the respondent has no confidence in their balance and 100 indicating that they are full confident that they can perform all items without a loss of balance. As such, higher values represent a better outcome. There are no sub-scales for this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Bastian, PhD, PT, Principal Investigator — Kennedy Krieger Institute and Johns Hopkins School of Medicine
Locations (1):
- Motion Analysis Lab in the Kennedy Krieger Institute, Baltimore, Maryland, United States